CLINICAL TRIAL: NCT00747838
Title: Surgical Treatment for Atrial Arrhythmia Registry (STAR Outcomes)
Brief Title: A Multicenter Data Registry for Outcomes From Surgical Treatment of Atrial Arrhythmias
Acronym: STAR
Status: Terminated | Type: Observational
Why Stopped: Low enrollment.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: STAR Outcomes
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Atrial Fibrillation
Keywords: Afib; Atrial Fibrillation; Maze; Mini-Maze
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Minimally Invasive Maze Procedure — Minimally Invasive Surgical Correction of Atrial Fibrillation.

SUMMARY:
Minimally invasive surgical treatment of atrial fibrillation is safe and effective at controlling atrial fibrillation. The fundamental goal of STAR Outcomes registry is to improve the understanding of the efficacy of surgical ablation intervention in the treatment of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with paroxysmal (intermittent) or persistent atrial fibrillation
2. > 18 years of age

Exclusion Criteria:

1. Patients unable to give adequate informed consent
2. Patients who are known to be pregnant, plan to become pregnant or are lactating
3. Inability to return for follow up
4. Patients who are prison inmates or institutionalized
5. Patients in an emergency state
6. Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with paroxysmal (intermittent) or persistent atrial fibrillation undergoing surgical correction.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Minimally invasive surgical treatment of atrial fibrillation is safe and effective at controlling atrial fibrillation | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Vigneshwar Kasirajan, MD, Principal Investigator — Virginia Commonwealth University; Kenneth Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Saini A, Hu YL, Kasirajan V, Han FT, Khan MZ, Wolfe L, Gunda S, Koneru JN, Ellenbogen KA. Long-term outcomes of minimally invasive surgical ablation for atrial fibrillation: A single-center experience. Heart Rhythm. 2017 Sep;14(9):1281-1288. doi: 10.1016/j.hrthm.2017.04.029. Epub 2017 Apr 22. PMID 28438723
- [Derived] Kasirajan V, Spradlin EA, Mormando TE, Medina AE, Ovadia P, Schwartzman DS, Gaines TE, Mumtaz MA, Downing SW, Ellenbogen KA. Minimally invasive surgery using bipolar radiofrequency energy is effective treatment for refractory atrial fibrillation. Ann Thorac Surg. 2012 May;93(5):1456-61. doi: 10.1016/j.athoracsur.2012.01.110. PMID 22541178
- [Derived] Kron J, Kasirajan V, Wood MA, Kowalski M, Han FT, Ellenbogen KA. Management of recurrent atrial arrhythmias after minimally invasive surgical pulmonary vein isolation and ganglionic plexi ablation for atrial fibrillation. Heart Rhythm. 2010 Apr;7(4):445-51. doi: 10.1016/j.hrthm.2009.12.008. Epub 2009 Dec 16. PMID 20156608